CLINICAL TRIAL: NCT05848856
Title: The Risk Informed Screening Registry (The RISC Registry)
Brief Title: The RISC Registry--Risk Informed Screening Registry
Acronym: RISC
Status: Not yet recruiting | Type: Observational
Sponsor: Precision Health Equity Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: RISC 1.01
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Risk; Cardiovascular Disease Risk; Cardiometabolic Risk; Diabetes
Keywords: Breast cancer; Diabetes; Obesity; Coronary artery disease; Risk; Prevention; Genetics; Social drivers of health; Personal risk adjusted screening plans
MeSH Terms: conditions — Diabetes Mellitus; Breast Neoplasms; Obesity; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Breast Cancer, Cardiometabolic, Cardiovascular Risk Screening and Follow up — Study of different types of risk-informed screening approaches and the measurement of patient compliance with screening recommendations based on different approaches to patient engagement

SUMMARY:
Chronic diseases such as heart disease, cancer, and diabetes are the leading causes of death and disability in the United States. Six in ten adults have one chronic disease; 4 in 10 have two or more. These are also leading drivers of the nation's $4.1 trillion in annual health care costs.

Cardiovascular disease is the number one cause of death for men and women, cancer is the second largest, with breast cancer being the second largest cause of death in women. Diabetes is the 8th highest cause of death for both men and women.

Routine screening, a focus on prevention, early detection, and patient engagement with proposed care plans, effective surveillance and follow up are some of the most effective ways to reduce the burden of chronic diseases across an individual's lifetime and at the population level.

Estimating dollar costs associated with non-compliance with screening and health management recommendations is complex and variable depending on the specific context, disease, and condition. But there is much evidence to indicate that a significant amount of these annual costs can be mitigated if compliance with health management recommendations increases, and health problems are prevented or detected early.

Access to screening and noncompliance with health management recommendations impact the entire population, but more disparities exist in racial and ethnic minorities and in the historically underserved for cancer, obesity, diabetes and cardiovascular disease.

The overall cost of these disparities in the U.S. has been estimated at around 1.24 trillion U.S. Dollars.

The RISC Registry seeks to pursue the intersection of breast cancer, metabolic, and cardiovascular risk in women and study the application of individualized multi-condition risk assessments, risk-informed or personalized screening, prevention and follow up care approaches in a broad cross section of patients. It pursues the hypothesis that these approaches accompanied by population appropriate methods of clinician and patient engagement may increase understanding and compliance with breast cancer, obesity, and metabolic/cardiovascular/cardiometabolic risk screening, surveillance and follow up recommendations by empowering women to make healthier choices.

In doing so, these methods may identify ways to address disparities in screening and patient care and ultimately promote early detection or even reversal of adverse health conditions, improve overall personal health, and reduce overall health care costs.

The primary focus is cancer, cardiovascular and metabolic health screening with a focus on utilization of Precision Screening. (Precision Screening attempts to separate those who will benefit from screening from those that may not, through use of information on disease risk.)

The study will start by focusing on women and risk for these diseases and health conditions.

DETAILED DESCRIPTION:
The RISC Registry (the "Registry") is a longitudinal observational database designed to capture health information that inform individualized disease risk and care plans in varied and diverse patient populations and study how that information impacts physician recommendations and patient compliance.

The Registry was designed by a board of Scientific Advisors who are active users of risk assessment tools, and risk-informed screening protocols, including physicians, nurses, and patient advocates. Technology professionals and site administrators were also consulted regarding optimizing the process of data collection and dissemination. The Registry uses widely accepted standards for risk and disease classifications, results, management, and validated quality-of-life measures.

The Registry is vendor-agnostic and product-agnostic. This study will make a special effort to reach women who have historically been underserved by recruiting patients broadly distributed across different socioeconomic groups, ethnicities and diverse geographic areas.

The RISC Registry will help determine the ongoing value of Precision Screening in different clinical patient populations, shape guidelines for screening and optimal patient management, and support improvements in Precision Health and Precision Medicine support technology.

Eligible subjects will be offered multi-disease personalized risk assessments and care plans at no charge to reduce cost as a barrier to screening.

ELIGIBILITY:
Inclusion Criteria:

* Female (Gender assigned at birth)
* Unaffected women (by breast cancer, diabetes or cardiovascular disease)
* Females who have been diagnosed with breast cancer, diabetes or cardiovascular disease
* Females who are presenting for cancer, metabolic health or cardiovascular screening
* Females presenting for mammography or other breast cancer screening procedures
* Females presenting for cholesterol, other blood tests aimed at metabolic and cardiovascular health screening, ECG's, EKG's or other noninvasive scans for the presence of or risk of heart disease
* Ages 18+
* Willing to sign a study consent form
* Willing to participate in PRO surveys
* Willing to use technology to participate in the study procedures, if and as needed
* Pregnant women may be included

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusive study of women who are seeking screening for breast cancer, cardiovascular disease and cardiometabolic risk
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2034-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease risks and issues identified during multi-condition risk assessment | Within 3 months
  Types of disease risks or issues identified by implementing a multi-condition risk assessment in a single patient.
Objective health measures within different population subgroups--blood pressure | Within 6 months
  Changes in an individual's blood pressure (both systolic and diastolic) tracked over time associated with different risk assessments, recommended care plans and patient engagement techniques, by different population subgroups. Could include data gathered from connected health devices used as part of the care plan and follow up.
Objective health measures within different population subgroups--BMI | Within 6 months
  Changes in an individual's BMI using combined height and weight measures, tracked over time, associated with different cardiovascular and breast cancer risk assessments, recommended care plans and patient engagement techniques, by different population subgroups.
Objective health measures within different population subgroups--HDL levels | Within 6 months
  Changes (increase or decrease) in an individual's HDL tracked over time associated with different risk assessments, recommended care plans and patient engagement techniques, by different population subgroups.
Objective health measures within different population subgroups-- abnormal germline genetic test results | Within 6 months
  Prevalence of abnormal germline genetic test results for cardiovascular and breast cancer disease risk, by different population sub groups
Number of subjects with newly diagnosed early stage cardiometabolic conditions and breast cancer | Within 6 months
  Early detection as measured by stage/extent of disease, linked to different risk assessments, care plans and patient engagement techniques, within different population subgroups.
Cancer health outcomes--imaging follow up | Within 1 year
  Short term cancer health outcomes using RECIST (Response Evaluation Criteria in Solid Tumors) to analyse how well treatment has worked as measured or detected by imaging results
Short and Long term cancer health outcomes--biospecimen tests | Within 1 year
  Short--within one year and longer term --within 5 years--cancer health outcomes using survival measure scales including Progression Free Survival (PFS) correlated with biospecimen tests that detect presence of disease.
Short and Long term cancer health outcomes--biospecimen tests | Within 1 year
  Short--within one year and longer term --within 5 years--cancer health outcomes using survival measure scales including Event Free Survival (EFS--complications and events the treatment was supposed to prevent) correlated with biospecimen tests that detect presence of disease.
PRO--Patient Reported Outcomes: Percent of time patient screening behaviors changed based on recommendations made by shared decision making with the clinician | Within 3 months
  Patient behavior correlated with recommendations evaluated by type of method of engagement and various social drivers of health (SDOH) using the PRAPARE survey (https://prapare.org/the-prapare-screening-tool/)
PRO--Patient Reported Outcomes: compliance with post screening recommendations | Within 3 months
  Patient compliance with recommendations evaluated by type of method of engagement and various social drivers of health (SDOH) as measured by using the PRAPARE survey (https://prapare.org/the-prapare-screening-tool/)
Clinician--Recommendations based on multi-condition risk assessments | Within 1 month
  Types of recommendations and percent (%) of time they change based on precision risk assessments

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, MD, Principal Investigator — Precision Health Equity Initiative
Locations (1):
- PHEI--Precision Health Equity Initiative, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
If PHEI does share participant data it will be after review by the PHEI Scientific Advisory Committee and all data will be de-indentified.